CLINICAL TRIAL: NCT01732107
Title: A Phase II Trial of Dovitinib in Bacillus Calmette-Guerin(BCG) Refractory Urothelial Carcinoma Patients With Tumor Fibroblast Growth Factor Receptor 3(FGFR3) Mutations or Over-expression: Hoosier Cancer Research Network GU12-157
Brief Title: Dovitinib in BCG Refractory Urothelial Carcinoma With FGFR3 Mutations or Over-expression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Development of dovitinib was stopped.
Sponsor: Noah Hahn, M.D. (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Noah Hahn, M.D., Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU12-157
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Bladder Cancer
Keywords: Dovitinib; FGFR3 Mutations; BCG-Refractory Urothelial Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dovitinib (Experimental): Dovitinib will be administered 500mg orally in a 5 days on, 2 days off dosing schedule.
  Interventions: Drug: Dovitinib

INTERVENTIONS:
Drug: Dovitinib — Dovitinib will be administered 500mg orally in a 5 days on, 2 days off dosing schedule. Day 12 assessments are intended to be performed on the last dosing day of the 2nd week in cycle 1 and cycle 2 and day 26 assessments are intended to be performed on the last dosing day of the 4th week in cycle 1 and cycle 2.

SUMMARY:
This trial will assess the 6-month complete response rate and toxicity profile of oral dovitinib therapy in BCG-refractory urothelial carcinoma patients with tumors with FGFR3 mutations or over-expression who are ineligible for or refusing cystectomy.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

* Dovitinib will be administered 500mg orally in a 5 days on, 2 days off dosing schedule. Day 12 assessments are intended to be performed on the last dosing day of the 2nd week in cycle 1 and cycle 2 and day 26 assessments are intended to be performed on the last dosing day of the 4th week in cycle 1 and cycle 2.
* Standard of Care: Cystoscopy with tumor biopsy, bladder biopsy, urine cytology
* Physician discretion: Anti-emetic medications and/or colony stimulating growth factors

ECOG performance status 0 - 2

Hematopoietic:

* White blood cell count (WBC) > 3.0 K/mm3
* Absolute neutrophil count (ANC) ≥ 1.5 K/mm3
* Platelets ≥ 100 K/mm3
* Hemoglobin (Hgb) ≥ 9 g/dL

Hepatic:

* Serum total bilirubin: ≤ 1.5 x Upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 3.0 x ULN

Renal:

* Serum creatinine ≤ 1.5 x ULN or serum creatinine > 1.5 - 3 x ULN if calculated creatinine clearance (CrCl) is ≥ 30 mL/min using the Cockcroft-Gault equation

Cardiovascular:

No impaired cardiac function or clinically significant cardiac diseases, including any of the following:

* History or presence of serious uncontrolled ventricular arrhythmias
* Clinically significant resting bradycardia
* LVEF assessed by 2-D echocardiogram (ECHO) < 50% or lower limit of normal (whichever is higher) or multiple gated acquisition scan (MUGA), < 45% or lower limit of normal (whichever is higher)
* Myocardial Infarction (MI), severe/unstable angina, Coronary Artery Bypass Graft (CABG), Congestive Heart Failure (CHF), Cerebrovascular Accident (CVA), Transient Ischemic Attack (TIA), Pulmonary Embolism (PE)within 6 months prior to starting study drug

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed early stage urothelial carcinoma of the bladder defined as Ta, T1, or Tis stage.
* Presence of either an FGFR3 mutation or FGFR3 over-expression within bladder tumor tissue.
* Documented BCG-refractory disease defined as failure to achieve a tumor free state after at least 2 prior induction courses of intravesical BCG therapy.
* Medically unfit to undergo cystectomy or electively choosing to forego cystectomy
* Patients who give a written informed consent obtained according to local guidelines

Exclusion Criteria:

* Patients with muscle-invasive (i.e. T2, T3, T4), locally advanced non-resectable, or metastatic urothelial carcinoma as assessed on baseline radiographic imaging obtained within 28 days prior to study registration.
* Patients with concurrent upper urinary tract (i.e. ureter, renal pelvis) non-invasive urothelial carcinoma.
* Patients with another primary malignancy within 3 years prior to starting study drug, with the exception of adequately treated in-situ carcinoma of the uterine cervix, clinically localized prostate cancer, biochemically relapsed non-metastatic prostate cancer (i.e., PSA only disease), or skin cancer (such as basal cell carcinoma, squamous cell carcinoma, or non-melanomatous skin cancer)
* Patients who have received the last administration of an anti-cancer therapy including chemotherapy, immunotherapy, and monoclonal antibodies ≤ 4 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy
* Patients who have received prior VEGFR-targeted or FGFR-targeted agents (i.e., sunitinib, pazopanib, sorafenib, bevacizumab, axitinib, etc.).
* Patients who have had radiotherapy ≤ 4 weeks prior to starting study drug, or who have not recovered from radiotherapy toxicities
* Patients who have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury ≤ 4 weeks prior to starting study drug, or patients who have had minor procedures (i.e., TURBT), percutaneous biopsies or placement of vascular access device ≤ 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury
* Uncontrolled hypertension defined by a systolic blood pressure (SBP) ≥ 160 mm Hg and/or d iastolic blood pressure (DBP) ≥ 100 mm Hg, with or without anti-hypertensive medication(s)
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of dovitinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory)
* Patients who are currently receiving anti-coagulation treatment with therapeutic doses of warfarin. Full-dose anti-coagulation with low molecular weight heparin is permitted.
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol
* Pregnant or breast-feeding women
* Women of child-bearing potential, who are biologically able to conceive, not employing two forms of highly effective contraception. Highly effective contraception must be used throughout the trial and up to 8 weeks after the last dose of study drug (e.g. male condom with spermicidal; diaphragm with spermicide; intra-uterine device). Oral, implantable, or injectable contraceptives that may be affected by cytochrome P450 interactions are not considered effective for this study. Women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test ≤ 14 days prior to starting study drug.
* Fertile males not willing to use contraception, as stated above
* Patients unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-03-06 (Actual); Study Completion 2017-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah Hahn, M.D., Study Chair — Hoosier Cancer Research Network
Locations (3):
- United States (3):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Johns Hopkins University: Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Fox Chase Cancer Center Extramural Research Program, Rockledge, Pennsylvania

REFERENCES:
- See also: Hoosier Oncology Group Website — http://www.hoosieroncologygroup.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dovitinib
Started | 13
Completed | 0
Not Completed | 13
Not completed — Adverse Event | 2
Not completed — Disease Progression | 8
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Dovitinib
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 70 [57 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Determine 6-Month Complete Response Rate
Description: The 6-month complete response rate is defined as the proportion of patients treated with dovitinib with no evidence of any remaining urothelial carcinoma tumors of any T-stage (including Tis) present within the bladder as assessed by standard of care cystoscopic examination with transurethral resection of bladder tumor (TURBT) and urine cytology performed at 6 months after initiation of study therapy.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Dovitinib
Number analyzed (Participants) | 13
percentage of participants | 8

2. Secondary Outcome: Determine 1-Year Relapse-Free Survival Rate
Description: The 1-year relapse free survival rate is defined as the proportion of patients treated with dovitinib with no evidence of any remaining urothelial carcinoma tumors at 12 months of follow-up.
Time Frame: 12 months
Population: Data for this outcome measure was neither collected or analyzed due to the early termination of the study.
Arm/Group | Dovitinib
Number analyzed (Participants) | 0

3. Secondary Outcome: Determine Rate of Progression to Muscle-Invasive Stage
Description: The rate of progression to muscle-invasive stage for dovitinib is defined as the proportion of patients with clinical or pathologic progression to muscle-invasive stages (i.e., T2-T4) at any time point on study.
Time Frame: 12 months
Population: Data for this outcome measure was neither collected or analyzed due to the early termination of the study.
Arm/Group | Dovitinib
Number analyzed (Participants) | 0

4. Secondary Outcome: Determine 3-Month and 6-Month Partial Response Rates
Description: The 3- and 6-month partial response rates are defined as the proportion of patients treated with persistent but reduced T-stage tumors on post-therapy TURBT (i.e., T1 ≥ Ta; T1+Tis ≥ T1).
Time Frame: 6 months
Population: Data for this outcome measure was neither collected or analyzed due to the early termination of the study.
Arm/Group | Dovitinib
Number analyzed (Participants) | 0

5. Secondary Outcome: Characterize Treatment-related Toxicity Rates
Description: Treatment-related toxicity rates will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0. All grade 3-4 adverse events and other adverse events occurring in more than 20% of patients are reported.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Dovitinib
Number analyzed (Participants) | 13
participants
  Fatigue (Grade 1) | 5
  Fatigue (Grade 2) | 4
  Fatigue (Grade 3) | 2
  Pain (Grade 1) | 6
  Pain (Grade 2) | 6
  Other Constitutional (Grade 1) | 3
  Other Constitutional (Grade 2) | 2
  Fall (Grade 3) | 1
  Hypertension (Grade 2) | 2
  Hypertension (Grade 3) | 2
  Headache (Grade 1) | 5
  Headache (Grade 2) | 1
  Headache (Grade 3) | 1
  Intracranial Hemmorage (Grade 3) | 1
  GERD (Grade 1) | 2
  GERD (Grade 2) | 3
  GERD (Grade 3) | 2
  Constipation (Grade 1) | 2
  Constipation (Grade 2) | 2
  Diarrhea (Grade 1) | 8
  Diarrhea (Grade 2) | 2
  Anorexia (Grade 1) | 4
  Anorexia (Grade 2) | 1
  Weight loss (Grade 1) | 4
  Dysgeusia (Grade 1) | 5
  Dysgeusia (Grade 2) | 2
  Nausea/Emesis (Grade 1) | 6
  Emesis (Grade 1) | 4
  Other gastrointestinal (Grade 1) | 2
  Other gastrointestinal (Grade 2) | 3
  Stomatitis (Grade 3) | 1
  Rash (Grade 1) | 4
  Rash (Grade 2) | 1
  Rash (Grade 3) | 1
  Hand-foot syndrome (Grade 1) | 2
  Hand-foot syndrome (Grade 2) | 1
  Dry mouth (Grade 1) | 4
  Other skin (Grade 1) | 6
  Other skin (Grade 2) | 2
  Bladder spasms (Grade 2) | 3
  Other urinary (Grade 1) | 7
  Other urinary (Grade 2) | 1
  Fever (Grade 1) | 4
  Infection (Grade 2) | 8
  Hoarseness (Grade 1) | 3
  Other pulmonary (Grade 1) | 4
  Other pulmonary (Grade 2) | 2
  Arthralgia/Myalgia (Grade 1) | 4
  Arthralgia/Myalgia (Grade 2) | 2
  Hypertriglyceridemia (Grade 1) | 1
  Hypertriglyceridemia (Grade 2) | 2
  Hypertriglyceridemia (Grade 3) | 1
  Hypertriglyceridemia (Grade 4) | 1
  Elevated alkaline phosphatase (Grade 1) | 2
  Elevated alkaline phosphatase (Grade 2) | 1
  Elevated GGT (Grade 2) | 1
  Elevated GGT (Grade 3) | 2
  Hypoalbuminemia (Grade 1) | 2
  Hypoalbuminemia (Grade 2) | 1
  Elevated lipase (Grade 3) | 2
  Other metabolic (Grade 1) | 6
  Anemia (Grade 1) | 4

6. Other Pre Specified Outcome: Characterize Pre- and Post-treatment Bladder Tumor FGFR Pathway Phosphorylation Changes.
Description: Pre- and post-treatment bladder tumor FGFR pathway phosphorylation changes will be assessed by bladder tumor tissue immunohistochemistry utilizing commercially available antibodies including, but not limited to, the following: fibroblast growth factor receptors (FGFR3, pFGFR3), vascular endothelial growth factor receptors (VEGFR2, pVEGFR2), fibroblast growth factor receptor substrates (2FRS2, pFRS2), extracellular signal-regulated kinases (ERK), phosphorylated extracellular signal-related kinase (pERK).
Time Frame: 12 months
Population: Data for this outcome measure was neither collected or analyzed due to the early termination of the study.
Arm/Group | Dovitinib
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Characterize Associations Between Pre-treatment Germline, FGFR Single-nucleotide Polymorphisms (SNPs) and Post-treatment 6-month Complete Response Rate and 1-year Relapse Free Survival Rate in Patients Treated With Dovitinib.
Description: Pre-treatment germline FGFR SNPs will be assessed by testing extracted Deoxyribonucleic acid (DNA) from patient peripheral blood mononuclear cells (PBMC's) (collected prior to initiating dovitinib therapy) with validated commercial probes.
Time Frame: 12 months
Population: Data for this outcome measure was neither collected or analyzed due to the early termination of the study.
Arm/Group | Dovitinib
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Characterize Pre- and Post-treatment VEGFR Pathway Phosphorylation Changes as Assessed by Bladder Tumor Tissue Immunohistochemistry.
Description: Pre- and post-treatment bladder tumor VEGFR pathway phosphorylation changes will be assessed by bladder tumor tissue immunohistochemistry utilizing commercially available antibodies including, but not limited to, the following: FGFR3, pFGFR3, VEGFR2, pVEGFR2, FRS2, pFRS2, ERK, pERK.
Time Frame: 12 months
Population: Data for this outcome measure was neither collected or analyzed due to the early termination of the study.
Arm/Group | Dovitinib
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Characterize Associations Between Pre-treatment Germline VEGFR SNPs and Post-treatment 6-month Complete Response Rate and 1-year Relapse Free Survival Rate in Patients Treated With Dovitinib.
Description: Pre-treatment germline VEGFR SNPs will be assessed by testing extracted DNA from patient PBMC's (collected prior to initiating dovitinib therapy) with validated commercial probes.
Time Frame: 12 months
Population: Data for this outcome measure was neither collected or analyzed due to the early termination of the study.
Arm/Group | Dovitinib
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Characterize Associations Between Post-treatment Hypertension, 6-month Complete Response Rate and 1-year Relapse Free Survival Rate in Patients Treated With Dovitinib.
Description: Hypertension will be defined as a systolic blood pressure (SBP) of > 140 mmHg or a diastolic blood pressure (DBP) of > 90 mm Hg recorded at any time after dovitinib therapy is initiated.
Time Frame: 12 months
Population: Data for this outcome measure was neither collected or analyzed due to the early termination of the study.
Arm/Group | Dovitinib
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Characterize Concordance Rates Between UC Patient Detected Tumor, Urine, and Circulating Free Plasma FGFR3 Mutations.
Description: Presence of FGFR3 mutations within patient free plasma will be assessed by polymerase chain reaction (PCR) amplification of the target regions and sequencing.
Time Frame: 12 months
Population: Data for this outcome measure was neither collected or analyzed due to the early termination of the study.
Arm/Group | Dovitinib
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Characterize Post-treatment Bladder Tissue Dovitinib Concentrations.
Description: Post-treatment bladder tissue dovitinib concentrations will be assessed by TURBT fresh frozen tissue obtained at the 3-month cystoscopy
Time Frame: 12 months
Population: 9 subjects had sufficient tissue available to measure dovitinib tissue concentration
Measure: Number; unit: nmol/L
Arm/Group | Dovitinib
Number analyzed (Participants) | 9
nmol/L
  Subject 2 | 1603
  Subject 3 | 159
  Subject 6 | 5813
  Subject 7 | 812
  Subject 8 | 726
  Subject 10 | 1135
  Subject 11 | 94
  Subject 12 | 2115
  Subject 13 | 2483

ADVERSE EVENTS:
Time Frame: Duration of participation of the treatment portion of the study, up to six cycles (6 Months).
Arm/Group | Dovitinib
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 3/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dovitinib (N=13)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
INTRACRANIAL HEMORRHAGE (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dovitinib (N=13)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (3)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (3)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 (5)
ANEMIA (Blood and lymphatic system disorders) | 6 (9)
ANOREXIA (Metabolism and nutrition disorders) | 5 (6)
ANXIETY (Psychiatric disorders) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4)
BLADDER SPASM (Renal and urinary disorders) | 4 (7)
BLURRED VISION (Eye disorders) | 1 (1)
BRUISING (Injury, poisoning and procedural complications) | 1 (1)
CARDIAC DISORDERS (Cardiac disorders) | 1 (1)
CATARACT (Eye disorders) | 1 (2)
CHEST PAIN - CARDIAC (Cardiac disorders) | 1 (2)
CHILLS (General disorders) | 1 (1)
CHOLESTEROL HIGH (Investigations) | 3 (6)
CONDUCTION DISORDER (Cardiac disorders) | 1 (1)
CONJUNCTIVITIS (Eye disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 6 (8)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CREATININE INCREASED (Investigations) | 1 (1)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 10 (15)
DIZZINESS (Nervous system disorders) | 2 (2)
DRY MOUTH (Gastrointestinal disorders) | 4 (4)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
DYSARTHRIA (Nervous system disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 7 (9)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
EAR AND LABYRINTH DISORDERS (Ear and labyrinth disorders) | 1 (1)
ESOPHAGEAL PAIN (Gastrointestinal disorders) | 1 (1)
EYE INFECTION (Infections and infestations) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (2)
FATIGUE (General disorders) | 11 (18)
FECAL INCONTINENCE (Gastrointestinal disorders) | 1 (1)
FEVER (General disorders) | 4 (7)
FLATULENCE (Gastrointestinal disorders) | 2 (2)
FLU LIKE SYMPTOMS (General disorders) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (3)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 1 (1)
GGT INCREASED (Investigations) | 3 (12)
HEADACHE (Nervous system disorders) | 8 (10)
HEARING IMPAIRED (Ear and labyrinth disorders) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 3 (3)
HEPATOBILIARY DISORDERS (Hepatobiliary disorders) | 1 (2)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 3 (3)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPERNATREMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 6 (27)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 5 (17)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPOKALEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 2 (4)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (1)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS (Injury, poisoning and procedural complications) | 1 (1)
INSOMNIA (Psychiatric disorders) | 2 (2)
INVESTIGATIONS (Investigations) | 1 (1)
LIPASE INCREASED (Investigations) | 3 (5)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1)
MALAISE (General disorders) | 1 (3)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER (Musculoskeletal and connective tissue disorders) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 6 (8)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (3)
ORAL PAIN (Gastrointestinal disorders) | 1 (2)
PAIN (General disorders) | 2 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
PAPULOPUSTULAR RASH (Infections and infestations) | 1 (1)
PARESTHESIA (Nervous system disorders) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 3 (3)
PLATELET COUNT DECREASED (Investigations) | 2 (2)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1)
PSYCHIATRIC DISORDERS (Psychiatric disorders) | 1 (1)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 3 (4)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 4 (4)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SERUM AMYLASE INCREASED (Investigations) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 2 (4)
SKIN HYPOPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN INFECTION (Infections and infestations) | 1 (1)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1)
STOMACH PAIN (Gastrointestinal disorders) | 2 (2)
TOOTHACHE (Gastrointestinal disorders) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1)
URINARY FREQUENCY (Renal and urinary disorders) | 6 (6)
URINARY TRACT INFECTION (Infections and infestations) | 4 (4)
URINARY TRACT PAIN (Renal and urinary disorders) | 1 (1)
URINARY URGENCY (Renal and urinary disorders) | 1 (1)
VOICE ALTERATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 4 (4)
WATERING EYES (Eye disorders) | 1 (1)
WEIGHT LOSS (Investigations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT01732107/Prot_SAP_000.pdf